CLINICAL TRIAL: NCT05430516
Title: Within Household Transmission of SARS-CoV-2 Infections, a Multicentre Prospective
Brief Title: Within Household Transmission of COVID-19 Infections
Acronym: VERDI
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Patricia Bruijning-Verhagen, Principal Investigator, UMC Utrecht
Other Study IDs: NL73581.041.20
Record Dates: First submitted 2022-03-17; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: SARS-CoV-2
Keywords: SARS-CoV-2; Omicron; Children; Household study; Tranmission

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Families: Patients with confirmed SARS-Cov-2 infection and their household members of all ages can be enrolled in the study, if at least one household member is a child age under 18.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
In the absence of a vaccine, the spread of SARS-CoV-2 can only be mitigated via non-pharmaceutical interventions that reduce the risks of forward transmission. Currently, European policymakers are implementing combinations of fierce pandemic control measures. However, there is substantial uncertainty on the transmission dynamics of SARS-CoV-2 and, consequently, the effect of each specific mitigation intervention as well as their joint impact on the pandemic evolution. Moreover, it is uncertain how and when the Public Health response should be modified once the pandemic starts to slow. There is an urgent need for data that can help to further unravel the key transmission characteristics of SARS-CoV-2 in the population. Household studies are, therefore, a useful approach to obtain insight into the main determinants of transmission and to derive estimates of transmission parameters. By fully characterizing the critical process of SARS-CoV-2 household transmission and how they vary by patient and household characteristics, infection dynamics in the population can be further elucidated.

Responding to SARS-CoV-2 effectively from a community care perspective will also require understanding the perceptions, beliefs, and actions taken by patients and the public.

A 'bottom-up' understating of such issues is critical to understand how best to design effective community strategies.

Rapid European COVID-19 Emergency Research response (RECOVER) is a project involving ten international partners that have been selected for funding by the European Union under the Horizon 2020 research framework. RECOVER responds to call topic SC1-PHE-CORONAVIRUS-2020: Advancing knowledge for the clinical and public health response to the SARS-CoV-2 epidemic and builds on many years of investment by the European Commission in clinical research preparedness for epidemic response. RECOVER will therefore provide a range of data and analytical results to guide the Public Health response, including the here described household transmission study.

Objective: Estimate key transmission parameters of SARS-CoV-2 in Europe from observing within household virus spread and seroconversion of household members and characterize the views and experiences of households regarding perceptions, practices regarding infection control, and impacts of imposed isolation measures.

ELIGIBILITY:
Inclusion Criteria:

* All members of the household or their legal guardians consent to participation
* All members of the household are willing to complete diaries and questionnaires for the duration of follow-up
* All members of the household are willing to, and capable of self-sampling nose-throat swabs, (a subset) saliva and capillary blood samples by finger. If parents/caretakers of young children are reluctant to take a blood sample from their child, this is no reason for exclusion.

Exclusion Criteria:

* Patients or household members who are unable to consent, or do not wish to provide informed consent.
* Children, pregnant women and patients lacking capacity will be included. Those lacking capacity to consent for themselves will be identified and consent will be sought from an appropriate consulted.
* Households who do not have daily access to a smartphone or tablet with internet connection, will be excluded, as follow-up of households requires the use of an interactive diary App.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Communty within the region of Utrecht
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Estimate key transmission parameters of SARS-CoV-2 in Europe from observing within household virus spread and seroconversion of household members through study completion, an average of 4 weeks. | Samples and data collected through study completion, an average of 4 weeks.
  Estimate key transmission parameters of SARS-CoV-2 in Europe from observing within household virus spread and seroconversion of household members. Including secondary attack rates and Transmission rate.

SECONDARY OUTCOMES:
Estimate the incubation period through study completion, an average of 4 weeks. | Samples and data collected through study completion, an average of 4 weeks.
  Infer from the data the transmission parameter incubation period.
Estimate the generation time through study completion, an average of 4 weeks. | Samples and data collected through study completion, an average of 4 weeks.
  Infer from the data the transmission parameter generation time.
Estimate the susceptibility through study completion, an average of 4 weeks. | Samples and data collected through study completion, an average of 4 weeks.
  Infer from the data susceptibility rate of different types of individuals. Calculated as follows: number of secondary cases / total number exposed.
Estimate the infectiousness through study completion, an average of 4 weeks. | Samples and data collected through study completion, an average of 4 weeks.
  Infer from the data infectiousness rate of different types of individuals. Calculated as follows: number of index cases with secondary transmission / total number of index cases.
Estimate the transmission through study completion, an average of 4 weeks. | Samples and data collected through study completion, an average of 4 weeks.
  Infer from the data the transmission rate of different types of households (e.g. number of household members, living conditions, sanitary facilities, pets) and behavioral characteristics.
Determine seroconversion rates and how this compares with virologically confirmed SARS-CoV-2 infections through study completion, an average of 4 weeks. | Samples and data collected through study completion, an average of 4 weeks.
  Determine seroconversion rates and how this compares with virologically confirmed SARS-CoV-2 infections

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Bruijning, MD PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided